CLINICAL TRIAL: NCT01220037
Title: The Effect of Age and Dietary Protein Intake on Myocellular Characteristics Following a Single Bout of Resistance Exercise in Healthy Men
Brief Title: Resistance Exercise in Healthy Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Lex Verdijk, Dr., Maastricht University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: MEC 09-3-080
Record Dates: First submitted 2010-10-07; First posted 2010-10-13 (Estimated); Last update posted 2013-10-28 (Estimated); Status verified 2013-10

CONDITIONS: Single Bout of Resistance Type Exercise; Standardized Diet

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Young regular diet (Experimental): During the time of the study this group will adhere to a standardized regular diet.
  Interventions: Behavioral: Adhere to a specific standardized diet for 4 days
- Young low protein diet (Experimental): During the time of the study this group will adhere to a standardized low protein diet.
  Interventions: Behavioral: Adhere to a specific standardized diet for 4 days
- Young high protein (Experimental): During the time of the study this group will adhere to a standardized high protein diet.
  Interventions: Behavioral: Adhere to a specific standardized diet for 4 days
- Elderly (Experimental): During the time of the study this group will adhere to a standardized high protein diet
  Interventions: Behavioral: Adhere to a specific standardized diet for 4 days

INTERVENTIONS:
Behavioral: Adhere to a specific standardized diet for 4 days — 24 h before the start of the intervention all subjects will adhere to a standardized diet for 4 days. Young subjects are randomly allocated to either a low protein diet, regular protein diet or high protein diet group. All elderly subjects will adhere to a regular protein diet comparable to the regular protein diet of the young subjects.

SUMMARY:
In the present study, the effects of age and dietary intake will be assessed on myocellular characteristics during 72 hours after a resistance type exercise session.

ELIGIBILITY:
Inclusion Criteria:

* healthy men between the ages of 18-30 or 70-85 years

Exclusion Criteria:

* Subjects with a recent history or current state of cardiovascular disease, COPD, Parkinson, rheumatoid arthritis, musculoskeletal/orthopaedic disorders, renal disorder, cognitive impairment.

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2010-04; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Muscle fiber myonuclear and stem cell content | baseline
Muscle fiber myonuclear and stem cell content | 12 hours after a single bout of resistance type exercise
Muscle fiber myonuclear and stem cell content | 24 hours after a single bout of resistance type exercise
Muscle fiber myonuclear and stem cell content | 48 hours after a single bout of resistance type exercise
Muscle fiber myonuclear and stem cell content | 72 hours after a single bout resistance type exercise

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University Medical Centre, Maastricht, Zuid Limburg, Netherlands

REFERENCES:
- [Derived] Snijders T, Verdijk LB, McKay BR, Smeets JS, van Kranenburg J, Groen BB, Parise G, Greenhaff P, van Loon LJ. Acute dietary protein intake restriction is associated with changes in myostatin expression after a single bout of resistance exercise in healthy young men. J Nutr. 2014 Feb;144(2):137-45. doi: 10.3945/jn.113.183996. Epub 2013 Dec 4. PMID 24306214